CLINICAL TRIAL: NCT03331536
Title: Skeletal Health in Bariatric Surgery Patients
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Society for Metabolic and Bariatric Surgery (Other)
Responsible Party: Principal Investigator, Jayleen M. Grams, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300000701
Record Dates: First submitted 2017-10-14; First posted 2017-11-06 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Bariatric Surgery; Osteoporosis; Fractures, Bone; Roux En-Y Gastric Bypass; Sleeve Gastrectomy; Menopause; Premenopause
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Roux en Y Gastric Bypass Pre-menopausal: Pre-menopausal women undergoing Roux en Y Gastric Bypass
  Interventions: Procedure: Roux en Y Gastric Bypass Pre-menopausal
- Roux en Y Gastric Bypass Post-menopausal: Post-menopausal women undergoing Roux en Y Gastric Bypass
  Interventions: Procedure: Roux en Y Gastric Bypass Post-menopausal
- Sleeve Gastrectomy Pre-menopausal: Pre-menopausal women undergoing Sleeve Gastrectomy
  Interventions: Procedure: Sleeve Gastrectomy Pre-menopausal
- Sleeve Gastrectomy Post-menopausal: Post-menopausal women undergoing Gastric Sleeve
  Interventions: Procedure: Sleeve Gastrectomy Post-menopausal

INTERVENTIONS:
Procedure: Roux en Y Gastric Bypass Pre-menopausal — The investigator aims to determine changes in skeletal health after Roux en Y Gastric Bypass in pre-menopausal women. Dual-energy x-ray absorptiometry (DXA) will be used to assess bone mineral density (BMD), including assessment for fracture risk (FRAX). Trabecular Bone Score (TBS) software will be used to adjust FRAX scores for bone microstructure and an enhanced fracture risk probability. Biochemical markers of bone metabolism and calcium homeostasis including serum bone alkaline phosphatase (BALP), osteocalcin, type 1 procollagen (P1NP), c-terminal telopeptide (CTX), calcium, albumin, parathyroid hormone (PTH), and 25-OH vitamin D will be assayed.
  Groups: Roux en Y Gastric Bypass Pre-menopausal
Procedure: Roux en Y Gastric Bypass Post-menopausal — The investigator aims to determine changes in skeletal health after Roux en Y Gastric Bypass in post-menopausal women. Dual-energy x-ray absorptiometry (DXA) will be used to assess bone mineral density (BMD), including assessment for fracture risk (FRAX). Trabecular Bone Score (TBS) software will be used to adjust FRAX scores for bone microstructure and an enhanced fracture risk probability. Biochemical markers of bone metabolism and calcium homeostasis including serum bone alkaline phosphatase (BALP), osteocalcin, type 1 procollagen (P1NP), c-terminal telopeptide (CTX), calcium, albumin, parathyroid hormone (PTH), and 25-OH vitamin D will be assayed.
  Groups: Roux en Y Gastric Bypass Post-menopausal
Procedure: Sleeve Gastrectomy Pre-menopausal — The investigator aims to determine changes in skeletal health after Sleeve Gastrectomy in pre-menopausal women. Dual-energy x-ray absorptiometry (DXA) will be used to assess bone mineral density (BMD), including assessment for fracture risk (FRAX). Trabecular Bone Score (TBS) software will be used to adjust FRAX scores for bone microstructure and an enhanced fracture risk probability. Biochemical markers of bone metabolism and calcium homeostasis including serum bone alkaline phosphatase (BALP), osteocalcin, type 1 procollagen (P1NP), c-terminal telopeptide (CTX), calcium, albumin, parathyroid hormone (PTH), and 25-OH vitamin D will be assayed.
  Groups: Sleeve Gastrectomy Pre-menopausal
Procedure: Sleeve Gastrectomy Post-menopausal — The investigator aims to determine changes in skeletal health after Sleeve Gastrectomy in post-menopausal women. Dual-energy x-ray absorptiometry (DXA) will be used to assess bone mineral density (BMD), including assessment for fracture risk (FRAX). Trabecular Bone Score (TBS) software will be used to adjust FRAX scores for bone microstructure and an enhanced fracture risk probability. Biochemical markers of bone metabolism and calcium homeostasis including serum bone alkaline phosphatase (BALP), osteocalcin, type 1 procollagen (P1NP), c-terminal telopeptide (CTX), calcium, albumin, parathyroid hormone (PTH), and 25-OH vitamin D will be assayed.
  Groups: Sleeve Gastrectomy Post-menopausal

SUMMARY:
The investigators propose a prospective cohort trial that will help to understand the impact of Roux-en-Y gastric bypass (RYGB) and sleeve gastrectomy (SG) in pre- and post-menopausal female bariatric patients.

DETAILED DESCRIPTION:
While highly effective both RYGB and SG may lead to increased bone resorption, decreased bone mass, and increased risk of some fractures. Very few studies have compared the effects of the RYGB and the SG on changes skeletal health and findings have been inconsistent. Furthermore, few studies have investigated the short- or long-term consequences of bariatric surgery on bone mineral density in pre- and post-menopausal women. To what extent and how bariatric surgery impacts the skeleton largely remains undetermined. Because estrogen is protective against osteoporosis and fractures, the majority of fractures occur in postmenopausal women. It is important that women have higher rates of obesity (38.3%) compared to men (34.3%) and that ≥67% of bariatric patients are women. Therefore, women may be at a significantly increased risk of developing osteoporosis. These data may help establish clinical guidelines to assess, maintain, and promote skeletal health in the preoperative and postoperative care of bariatric patients; and it may help to determine the appropriate bariatric procedure for women at risk of osteoporosis and fractures.

ELIGIBILITY:
Inclusion Criteria:

* Adult females ≥ 19 years scheduled to undergo bariatric surgery (Roux en Y Gastric Bypass or Gastric Sleeve Surgery)
* Class II (BMI 35-39.9 kg/m2).
* Class III obesity (BMI ≥ 40 kg/m2).
* Scheduled to undergo bariatric surgery with the ability to provide informed consent.

Exclusion Criteria:

* Patients with a history of thyroid disorders, thyroidectomy and levothyroxine use.
* Patients with a history of known osteoporosis, steroid-induced osteoporosis, current or previous use of medications for osteoporosis.
* Patients with a history of gastrointestinal malabsorption.
* Patients with a history of renal diseases.
* Patients with a history of current or previous use of corticosteroids.
* Patients who have used tobacco products within a year of study enrollment.
* Patients with surgically-induced menopause e.g. bilateral salpingo-oophorectomy.
* Patients with a history of breast cancer, who have had or are currently on hormonal therapy or anti-hormonal therapy.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female bariatric surgery population scheduled to undergo Roux en Y Gastric Bypass or Gastric Sleeve Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2020-08-02 (Actual); Study Completion 2020-08-02 (Actual)

PRIMARY OUTCOMES:
Determine and quantify changes in bone mineral density after bariatric surgery (Roux en Y vs. Gastric Sleeve) in pre- and post-menopausal women. | Baseline
  Dual-energy x-ray absorptiometry (DXA) will be used to assess bone mineral density, BMD (in g/cm2) of the lumbar spine (L1-L4), total hip, femoral neck, distal radius, sub-total whole body (excluding only the head), and whole body. T scores will be evaluated and Z scores will be evaluated. T-scores between +1 and -1 is considered normal or healthy, T-scores between -1 and -2.5 indicates that you have low bone mass, although not low enough to be diagnosed with osteoporosis, T-scores of -2.5 or lower indicates that you have osteoporosis. For premenopausal women under the age of 50, the Z-score is used for diagnosis. Using the criteria defined by the International Society for Clinical Densitometry: If the Z-score is -2.0 or lower, the result will be below the expected range for age. If the Z score is above -2.0, the result is will be defined as within the expected range for age.
Determine and quantify changes in bone mineral density after bariatric surgery (Roux en Y vs. Gastric Sleeve) in pre- and post-menopausal women. | Baseline to 12 months
  Dual-energy x-ray absorptiometry (DXA) will be used to assess bone mineral density, BMD (in g/cm2) of the lumbar spine (L1-L4), total hip, femoral neck, distal radius, sub-total whole body (excluding only the head), and whole body. T scores will be evaluated and Z scores will be evaluated. T-scores between +1 and -1 is considered normal or healthy, T-scores between -1 and -2.5 indicates that you have low bone mass, although not low enough to be diagnosed with osteoporosis, T-scores of -2.5 or lower indicates that you have osteoporosis. For premenopausal women under the age of 50, the Z-score is used for diagnosis. Using the criteria defined by the International Society for Clinical Densitometry: If the Z-score is -2.0 or lower, the result will be below the expected range for age. If the Z score is above -2.0, the result is will be defined as within the expected range for age.
Determine and quantify changes in bone mineral density after bariatric surgery (Roux en Y vs. Gastric Sleeve) in pre- and post-menopausal women. | Baseline to 24 months
  Dual-energy x-ray absorptiometry (DXA) will be used to assess bone mineral density, BMD (in g/cm2) of the lumbar spine (L1-L4), total hip, femoral neck, distal radius, sub-total whole body (excluding only the head), and whole body. T scores will be evaluated and Z scores will be evaluated. T-scores between +1 and -1 is considered normal or healthy, T-scores between -1 and -2.5 indicates that you have low bone mass, although not low enough to be diagnosed with osteoporosis, T-scores of -2.5 or lower indicates that you have osteoporosis. For premenopausal women under the age of 50, the Z-score is used for diagnosis. Using the criteria defined by the International Society for Clinical Densitometry: If the Z-score is -2.0 or lower, the result will be below the expected range for age. If the Z score is above -2.0, the result is will be defined as within the expected range for age.
Fracture risk assessment in pre and post-menopausal women undergoing bariatric surgery (Roux en Y vs. Gastric Sleeve). | Baseline
  Assessment of fracture risk using the WHO Fracture Risk Assessment Tool (FRAX) will be used to assess the 10-year fracture risk probability (in %)
Fracture risk assessment in pre and post-menopausal women undergoing bariatric surgery (Roux en Y vs. Gastric Sleeve). | Baseline to 12 months
  Assessment of fracture risk using the WHO Fracture Risk Assessment Tool (FRAX) will be used to assess the 10-year fracture risk probability (in %)
Fracture risk assessment in pre and post-menopausal women undergoing bariatric surgery (Roux en Y vs. Gastric Sleeve). | Baseline to 24 months
  Assessment of fracture risk using the WHO Fracture Risk Assessment Tool (FRAX) will be used to assess the 10-year fracture risk probability (in %)
TBS adjustment of FRAX scores for an enhanced fracture risk probability in pre and post-menopausal women undergoing bariatric surgery (Roux en Y vs. Gastric Sleeve). | Baseline
  The Trabecular Bone Score (TBS) is derived from the texture of the DXA image and has been shown to be related to fracture risk. Trabecular Bone Score (TBS) software will be used to adjust fracture risk (FRAX) scores to obtain TBS scores (in gradient risk). FRAX adjusted TBS scores (in gradient of risk) ranges from 1.1% -1.9% coefficient of variation (C.V.)
TBS adjustment of FRAX scores for an enhanced fracture risk probability in pre and post-menopausal women undergoing bariatric surgery (Roux en Y vs. Gastric Sleeve). | Change from baseline to 12 months
  The Trabecular Bone Score (TBS) is derived from the texture of the DXA image and has been shown to be related to fracture risk. Trabecular Bone Score (TBS) software will be used to adjust fracture risk (FRAX) scores to obtain TBS scores (in gradient risk). FRAX adjusted TBS scores (in gradient of risk) ranges from 1.1% -1.9% coefficient of variation (C.V.)
TBS adjustment of FRAX scores for an enhanced fracture risk probability in pre and post-menopausal women undergoing bariatric surgery (Roux en Y vs. Gastric Sleeve). | Change from baseline to 24 months
  The Trabecular Bone Score (TBS) is derived from the texture of the DXA image and has been shown to be related to fracture risk. Trabecular Bone Score (TBS) software will be used to adjust fracture risk (FRAX) scores to obtain TBS scores (in gradient risk). FRAX adjusted TBS scores (in gradient of risk) ranges from 1.1% -1.9% coefficient of variation (C.V.)
TBS assessment of bone microstructure in pre and post-menopausal women undergoing bariatric surgery (Roux en Y vs. Gastric Sleeve). | Baseline
  The Trabecular Bone Score (TBS) is derived from the texture of the DXA image and has been shown to be related to bone microarchitecture. Trabecular Bone Score (TBS) software will be used to assess bone microstructure. TBS ≤1.2 defines degraded microarchitecture, TBS between 1.20 and 1.35 is partially degraded microarchitecture, and TBS ≥1.35 is considered normal.
TBS assessment of bone microstructure in pre and post-menopausal women undergoing bariatric surgery (Roux en Y vs. Gastric Sleeve). | Change from baseline to 12 months
  The Trabecular Bone Score (TBS) is derived from the texture of the DXA image and has been shown to be related to bone microarchitecture. Trabecular Bone Score (TBS) software will be used to assess bone microstructure. TBS ≤1.2 defines degraded microarchitecture, TBS between 1.20 and 1.35 is partially degraded microarchitecture, and TBS ≥1.35 is considered normal.
TBS assessment of bone microstructure in pre and post-menopausal women undergoing bariatric surgery (Roux en Y vs. Gastric Sleeve). | Change from baseline to 24 months
  The Trabecular Bone Score (TBS) is derived from the texture of the DXA image and has been shown to be related to bone microarchitecture. Trabecular Bone Score (TBS) software will be used to assess bone microstructure. TBS ≤1.2 defines degraded microarchitecture, TBS between 1.20 and 1.35 is partially degraded microarchitecture, and TBS ≥1.35 is considered normal.

SECONDARY OUTCOMES:
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline
  Serum bone alkaline phosphatase (BALP in U/L) will be assayed
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 6 months
  Serum bone alkaline phosphatase (BALP in U/L) will be assayed
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 12 months
  Serum bone alkaline phosphatase (BALP in U/L) will be assayed
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 24 months
  Serum bone alkaline phosphatase (BALP in U/L) will be assayed
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline
  Osteocalcin (in ng/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 6 months
  Osteocalcin (in ng/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 12 months
  Osteocalcin (in ng/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 24 months
  Osteocalcin (in ng/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline
  Type 1 procollagen (P1NP, in mcg/L) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 6 months
  Type 1 procollagen (P1NP, in mcg/L) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 12 months
  Type 1 procollagen (P1NP, in mcg/L) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 24 months
  Type 1 procollagen (P1NP, in mcg/L) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline
  C-terminal telopeptide (CTX, in pg/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 6 months
  C-terminal telopeptide (CTX, in pg/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 12 months
  C-terminal telopeptide (CTX, in pg/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 24 months
  C-terminal telopeptide (CTX, in pg/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline
  Calcium (in mg/dL), albumin (in, g/dL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 6 months
  Calcium (in mg/dL), albumin (in, g/dL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 12 months
  Calcium (in mg/dL), albumin (in, g/dL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 24 months
  Calcium (in mg/dL), albumin (in, g/dL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline
  Parathyroid hormone (PTH, in pg/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 6 months
  Parathyroid hormone (PTH, in pg/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 12 months
  Parathyroid hormone (PTH, in pg/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 24 months
  Parathyroid hormone (PTH, in pg/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline
  25-OH vitamin D (in ng/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 6 months
  25-OH vitamin D (in ng/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 12 months
  25-OH vitamin D (in ng/mL) will be assayed.
Determine and quantify changes in biochemical markers of bone metabolism and calcium homeostasis. | Baseline to 24 months
  25-OH vitamin D (in ng/mL) will be assayed.

CONTACTS AND LOCATIONS:
Overall Officials: Jayleen G Grams, MD,PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Kirklin Clinic Digestive Health Center, Birmingham, Alabama, United States